CLINICAL TRIAL: NCT02533427
Title: A Phase 1, Open-Label, Drug Interaction Study Evaluating the Effect of Sofosbuvir/Velpatasvir/GS-9857 Fixed-Dose Combination on the Pharmacokinetics of a Representative Hormonal Contraceptive Medication, Norgestimate/Ethinyl Estradiol
Brief Title: Study to Evaluate Effect of Sofosbuvir/Velpatasvir/GS-9857 Fixed-Dose Combination on the Pharmacokinetics of a Representative Hormonal Contraceptive Medication, Norgestimate/Ethinyl Estradiol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-367-1909
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination; voxilaprevir; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOF/VEL/VOX + VOX (Experimental): Part A: Participants without a documented history of taking norgestimate/ethinyl estradiol for at least one menstrual cycle will receive norgestimate/ethinyl estradiol. Participants with a documented history of taking norgestimate/ethinyl estradiol may enroll directly into Part B of the study.
  Part B: Participants will continue taking norgestimate/ethinyl estradiol for the remainder of the study and will receive SOF/VEL/VOX FDC plus VOX.
  Interventions: Drug: SOF/VEL/VOX; Drug: VOX; Drug: Norgestimate/ethinyl estradiol

INTERVENTIONS:
Drug: SOF/VEL/VOX — 400/100/100 mg FDC tablet administered orally once daily
  Other Names: Epclusa®
Drug: VOX — 100 mg tablet administered orally once daily
  Other Names: GS-9857
Drug: Norgestimate/ethinyl estradiol — Norgestimate 0.180 mg/0.215 mg/0.25 mg/ethinyl estradiol 0.025 mg tablet administered orally once daily according to the package insert
  Other Names: Ortho-Tri-Cyclen® Lo

SUMMARY:
This study will evaluate the effect of sofosbuvir (SOF)/velpatasvir (VEL)/voxilaprevir (VOX) fixed-dose combination (FDC) + voxilaprevir on the pharmacokinetics (PK) of a representative hormonal contraceptive medication, norgestimate/ethinyl estradiol (Ortho Tri-Cyclen® Lo (OC)) and will assess the effect of norgestimate/ethinyl estradiol on the PK of SOF/VEL/VOX+VOX.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female
* Must have a calculated body mass index (BMI) ≥ 19.0 and ≤ 30.0 kg/m^2 at screening
* Must have a negative serum pregnancy test at screening and urine pregnancy test at Day -1
* Be willing and able to comply with all study requirements.

Exclusion Criteria:

* Lactating female
* Have a history of any of the following:

  * Significant drug sensitivity or drug allergy (such as anaphylaxis or hepatoxicity)
  * Known hypersensitivity to the study drugs, the metabolites or formulation excipients
* Believed, by the study investigator, to be inappropriate for study participation for any reason

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2016-03-18 (Actual); Study Completion 2016-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a study site in New Zealand. The first participant was screened on 29 October 2015. The last study visit occurred on 18 March 2016.
Pre-assignment Details: 15 participants were screened.
Groups:
- NGM/EE + SOF/VEL/VOX + VOX (Part A and Part B): Part A: Participants without a documented history of taking norgestimate/ethinyl estradiol (NGM/EE) for at least one menstrual cycle received NGM 0.180 mg/0.215 mg/0.25 mg/ EE 0.025 mg tablet orally once daily for one cycle (cycle=28 days).
  Part B: Participants continued NGM/EE through Cycle 1 and 2 received sofosbuvir (SOF)/velpatasvir (VEL)/voxilaprevir (VOX) fixed dose combination (FDC) 400/100/100 mg tablet + VOX 100 mg tablet orally once daily during cycle 2 (cycle=28 days).
Period: Overall Study
Arm/Group | NGM/EE + SOF/VEL/VOX + VOX (Part A and Part B)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all enrolled participants who took at least 1 dose of study drug.
Arm/Group | NGM/EE + SOF/VEL/VOX + VOX (Part A and Part B)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of Norelgestromin
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Cycle 1,Study Day 14: Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose; Cycle 2,Study Day 42: Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose
Population: The PK Analysis Set included all enrolled participants who took at least 1 dose of study drug and had at least 1 non-missing postdose plasma concentration value reported.
Measure: Mean (Standard Deviation); unit: hours*picogram/milliliter (h*pg/mL)
Groups:
- Part A: NGM/EE: Participants received NGM 0.180 mg/0.215 mg/0.25 mg/ EE 0.025 mg tablet orally once daily for cycle 1 (cycle = 28 days).
- Part B: NGM/EE + SOF/VEL/VOX + VOX: Participants received NGM 0.180 mg/0.215 mg/0.25 mg/ EE 0.025 mg + sofosbuvir (SOF)/velpatasvir (VEL)/voxilaprevir (VOX) FDC 400/100/100 mg tablet + VOX 100 mg tablet orally once daily during cycle 2 (cycle = 28 days).
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
hours*picogram/milliliter (h*pg/mL) | 13757.4 (2478.44) | 14690.4 (2116.43)
Statistical Analysis 1: Comparison: Part A: NGM/EE vs Part B: NGM/EE + SOF/VEL/VOX + VOX; Norelgestromin Part B/Part A; Test type: Other; % Geometric Least Square Mean(GLSM)Ratio = 107.36, 90% CI 2-sided [103.19 to 111.69] — Test/Reference: Norelgestromin Part B/Part A

2. Primary Outcome: PK Parameter: AUCtau of Norgestrel
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: hours*nanogram/milliliter (h*ng/mL)
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
hours*nanogram/milliliter (h*ng/mL) | 41.1 (11.05) | 47.3 (13.19)
Statistical Analysis 1: Comparison: Part A: NGM/EE vs Part B: NGM/EE + SOF/VEL/VOX + VOX; Norgestrel Part B/Part A; Test type: Other; % GLSM Ratio = 115.14, 90% CI 2-sided [106.49 to 124.50] — Test/Reference: Norgestrel Part B/Part A

3. Primary Outcome: PK Parameter: AUCtau of Ethinyl Estradiol
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
h*pg/mL | 835.2 (367.17) | 871.4 (355.33)
Statistical Analysis 1: Comparison: Part A: NGM/EE vs Part B: NGM/EE + SOF/VEL/VOX + VOX; Ethinyl estradiol Part B/Part A; Test type: Other; % GLSM Ratio = 105.43, 90% CI 2-sided [96.95 to 114.66] — Test/Reference: Ethinyl estradiol Part B/Part A

4. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of Norgestimate
Description: as for outcome 1
Time Frame: Cycle 1,Study Day 14:Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose; Cycle 2,Study Day 42: Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 1 | 4
h*ng/mL | 0.2 (NA) — Standard deviation was not calculated as data was available for only one participant. | 0.5 (0.48)
Statistical Analysis 1: Comparison: Part A: NGM/EE vs Part B: NGM/EE + SOF/VEL/VOX + VOX; Norgestimate Part B/Part A; Test type: Other; % GLSM Ratio = 248.89, 90% CI 2-sided [33.11 to 1870.81] — Test/Reference: Norgestimate Part B/Part A

5. Primary Outcome: PK Parameter: Cmax of Norelgestromin
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
pg/mL | 1080.9 (221.11) | 1162.2 (209.53)
Statistical Analysis 1: Comparison: Part A: NGM/EE vs Part B: NGM/EE + SOF/VEL/VOX + VOX; Norelgestromin Part B/Part A; Test type: Other; % GLSM Ratio = 107.71, 90% CI 2-sided [97.78 to 118.65] — Test/Reference: Norelgestromin Part B/Part A

6. Primary Outcome: PK Parameter: Cmax of Norgestrel
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
ng/mL | 2.0 (0.52) | 2.3 (0.61)
Statistical Analysis 1: Comparison: Part A: NGM/EE vs Part B: NGM/EE + SOF/VEL/VOX + VOX; Norgestrel Part B/Part A; Test type: Other; % GLSM Ratio = 115.02, 90% CI 2-sided [108.12 to 122.37] — Test/Reference: Norgestrel Part B/Part A

7. Primary Outcome: PK Parameter: Cmax of Ethinyl Estradiol
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
pg/mL | 68.4 (31.06) | 80.6 (28.44)
Statistical Analysis 1: Comparison: Part A: NGM/EE vs Part B: NGM/EE + SOF/VEL/VOX + VOX; Ethinyl estradiol Part B/Part A; Test type: Other; % GLSM Ratio = 121.06, 90% CI 2-sided [106.10 to 138.12] — Test/Reference: Ethinyl estradiol Part B/Part A

8. Primary Outcome: PK Parameter: Cmax of Norgestimate
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
ng/mL | 0.0 (0.04) | 0.1 (0.05)
Statistical Analysis 1: Comparison: Part A: NGM/EE vs Part B: NGM/EE + SOF/VEL/VOX + VOX; Norgestimate Part B/Part A; Test type: Other; % GLSM Ratio = 112.11, 90% CI 2-sided [87.19 to 144.14] — Test/Reference: Norgestimate Part B/Part A

9. Primary Outcome: PK Parameter: Ctau of Norelgestromin
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Part A:Cycle 1,Study Day 14:Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose; Part B:Cycle 2,Study Day 42:Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
picogram/milliliter (pg/mL) | 364.1 (76.74) | 413.9 (73.78)
Statistical Analysis 1: Comparison: Part A: NGM/EE vs Part B: NGM/EE + SOF/VEL/VOX + VOX; Norelgestromin Part B/Part A; Test type: Other; % GLSM Ratio = 114.19, 90% CI 2-sided [107.40 to 121.39] — Test/Reference: Norelgestromin Part B/Part A

10. Primary Outcome: PK Parameter: Ctau of Norgestrel
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
nanogram/milliliter (ng/mL) | 1.5 (0.37) | 1.8 (0.55)
Statistical Analysis 1: Comparison: Part A: NGM/EE vs Part B: NGM/EE + SOF/VEL/VOX + VOX; Norgestrel Part B/Part A; Test type: Other; % GLSM Ratio = 121.62, 90% CI 2-sided [110.85 to 133.44] — Test/Reference: Norgestrel Part B/Part A

11. Primary Outcome: PK Parameter: Ctau of Ethinyl Estradiol
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
pg/mL | 19.7 (10.82) | 18.2 (10.39)
Statistical Analysis 1: Comparison: Part A: NGM/EE vs Part B: NGM/EE + SOF/VEL/VOX + VOX; Ethinyl estradiol Part B/Part A; Test type: Other; % GLSM Ratio = 92.86, 90% CI 2-sided [82.55 to 104.45] — Test/Reference: Ethinyl estradiol Part B/Part A

12. Primary Outcome: PK Parameter: Ctau of Norgestimate
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Cycle 1,Study Day 14: Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose;Cycle 2,Study Day 42: Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 6 | 3
ng/mL | 0.0 (0.00) | 0.0 (0.00)

13. Secondary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events
Time Frame: First dose date up to the last dose date (maximum: 84 days) plus 10 days
Population: The Safety Analysis Set included all enrolled participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
percentage of participants | 66.7 | 93.3

14. Secondary Outcome: Percentage of Participants Who Experienced Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each participant. Grade 1: mild; Grade 2: moderate;Grade 3: severe or medically significant but not immediately life-threatening; Grade 4: life-threatening consequences.
Time Frame: First dose date up to the last dose date (maximum: 84 days) plus 10 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
percentage of participants
  Grade 1 | 60.0 | 53.3
  Grade 2 | 13.3 | 6.7
  Grade 3 | 13.3 | 0.0
  Grade 4 | 0.0 | 0.0

15. Secondary Outcome: PK Parameter: Tmax of Norelgestromin, Norgestrel, Ethinyl Estradiol, and Norgestimate
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set with available were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
hours
  Norelgestromin | 3.00 [2.00 to 4.00] | 3.00 [1.50 to 4.00]
  Norgestrel | 4.00 [2.50 to 8.00] | 4.00 [2.50 to 6.00]
  Ethinyl Estradiol | 3.00 [1.50 to 3.00] | 2.00 [1.50 to 3.13]
  Norgestimate: number analyzed (Participants) | 9 | 12
  Norgestimate | 1.50 [1.00 to 1.50] | 1.50 [1.25 to 3.00]

16. Secondary Outcome: PK Parameter: Tlast of Norelgestromin, Norgestrel, Ethinyl Estradiol, and Norgestimate
Description: Tlast is defined as the time (observed time point) of Clast.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
hours
  Norelgestromin | 24.00 [24.00 to 24.00] | 24.00 [24.00 to 24.00]
  Norgestrel | 24.00 [24.00 to 24.00] | 24.00 [24.00 to 24.00]
  Ethinyl Estradiol | 24.00 [24.00 to 24.00] | 24.00 [24.00 to 24.00]
  Norgestimate: number analyzed (Participants) | 9 | 12
  Norgestimate | 1.50 [1.50 to 2.00] | 2.75 [2.00 to 3.00]

17. Secondary Outcome: PK Parameter: λz of Norelgestromin, Norgestrel, Ethinyl Estradiol, and Norgestimate
Description: λz is defined as the terminal elimination rate constant, estimated by linear regression of the terminal elimination phase of the log plasma concentration of drug versus time curve of the drug.
Time Frame: Cycle 1,Study Day 14: Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose; Cycle 2,Study Day 42:Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 1/hours (1/h)
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
1/hours (1/h)
  Norelgestromin | 0.035 (0.0095) | 0.025 (0.0084)
  Norgestrel: number analyzed (Participants) | 15 | 11
  Norgestrel | 0.016 (0.0081) | 0.012 (0.0039)
  Ethinyl Estradiol | 0.053 (0.0230) | 0.059 (0.0186)
  Norgestimate: number analyzed (Participants) | 1 | 4
  Norgestimate | 0.674 (NA) — Standard deviation was not calculated as data was available for only one participant. | 0.392 (0.3674)

18. Secondary Outcome: PK Parameter: t1/2 of Norelgestromin, Norgestrel, Ethinyl Estradiol, and Norgestimate
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
hours
  Norelgestromin | 18.91 [17.08 to 23.42] | 28.95 [21.90 to 36.02]
  Norgestrel: number analyzed (Participants) | 15 | 11
  Norgestrel | 33.76 [30.76 to 78.76] | 57.42 [49.41 to 82.93]
  Ethinyl Estradiol | 13.68 [10.01 to 21.06] | 10.78 [9.48 to 15.67]
  Norgestimate: number analyzed (Participants) | 1 | 4
  Norgestimate | 1.03 [1.03 to 1.03] | 2.30 [1.49 to 7.86]

19. Secondary Outcome: PK Parameter: CLss/F Ethinyl Estradiol, and Norgestimate
Description: CLss/F is defined as the apparent steady state oral clearance following administration of the drug.
Time Frame: \Cycle 1,Study Day 14: Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose; Cycle 2,Study Day 42: Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: milliliter/hour (mL/h)
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15 | 15
milliliter/hour (mL/h)
  Ethinyl Estradiol | 34226.8 (12691.91) | 32000.0 (9530.52)
  Norgestimate: number analyzed (Participants) | 1 | 4
  Norgestimate | 1285855.5 (NA) — Standard deviation was not calculated as data was available for only one participant. | 617498.8 (350620.05)

20. Secondary Outcome: PK Parameter: Cmax of Sofosbuvir (SOF), SOF Metabolites (GS-566500 and GS-331007), Velpatasvir (VEL), and Voxilaprevir (VOX)
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Cycle 2, Study Day 42: Predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours postdose
Population: Participants in the PK Analysis Set who were enrolled in Part B and received NGM+ SOV/VEL/VOX + VOX were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15
ng/mL
  SOF | 967.6 (322.20)
  GS-566500 | 491.1 (107.66)
  GS-331007 | 979.4 (119.43)
  VEL | 853.3 (161.60)
  VOX | 512.4 (171.71)

21. Secondary Outcome: PK Parameter: Tmax of SOF, SOF Metabolites (GS-566500 and GS-331007), VEL, and VOX
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: as for outcome 20
Population: Participants in the PK Analysis Set who were enrolled in Part B and received NGM+ SOV/VEL/VOX + VOX were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15
hours
  SOF | 2.50 [1.00 to 3.00]
  GS-566500 | 4.00 [3.00 to 4.00]
  GS-331007 | 4.00 [4.00 to 6.00]
  VEL | 4.00 [4.00 to 6.00]
  VOX | 6.00 [4.00 to 6.02]

22. Secondary Outcome: PK Parameter: Tlast of SOF, SOF Metabolites (GS-566500 and GS-331007), VEL, and VOX
Description: Tlast is defined as the time (observed time point) of Clast.
Time Frame: as for outcome 20
Population: Participants in the PK Analysis Set who were enrolled in Part B and received NGM+ SOV/VEL/VOX + VOX were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15
hours
  SOF | 6.00 [6.00 to 8.00]
  GS-566500 | 16.00 [16.00 to 20.00]
  GS-331007 | 24.00 [24.00 to 24.00]
  VEL | 24.00 [24.00 to 24.00]
  VOX | 24.00 [24.00 to 24.00]

23. Secondary Outcome: PK Parameter: Ctau of SOF Metabolites (GS-566500 and GS-331007), VEL, and VOX
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: as for outcome 20
Population: Participants in the PK Analysis Set who were enrolled in Part B and received NGM+ SOV/VEL/VOX + VOX were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15
ng/mL
  GS-566500: number analyzed (Participants) | 1
  GS-566500 | 10.6 (NA) — Standard deviation was not calculated as data was available for only one participant.
  GS-331007 | 323.1 (67.24)
  VEL | 154.6 (46.71)
  VOX | 56.1 (59.02)

24. Secondary Outcome: PK Parameter: λz of SOF, SOF Metabolites (GS-566500 and GS-331007), VEL, and VOX
Description: as for outcome 17
Time Frame: as for outcome 20
Population: Participants in the PK Analysis Set who were enrolled in Part B and received NGM+ SOV/VEL/VOX + VOX were analyzed.
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15
1/h
  SOF | 1.160 (0.4753)
  GS-566500 | 0.247 (0.0247)
  GS-331007 | 0.020 (0.0091)
  VEL | 0.037 (0.0103)
  VOX | 0.077 (0.0277)

25. Secondary Outcome: PK Parameter: AUCtau of SOF, SOF Metabolites (GS-566500 and GS-331007), VEL, and VOX
Description: as for outcome 1
Time Frame: as for outcome 20
Population: Participants in the PK Analysis Set who were enrolled in Part B and received NGM+ SOV/VEL/VOX + VOX were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15
h*ng/mL
  SOF | 1997.2 (802.99)
  GS-566500 | 2769.3 (446.51)
  GS-331007 | 12098.9 (1929.14)
  VEL | 8226.3 (2056.25)
  VOX | 3857.9 (1216.12)

26. Secondary Outcome: PK Parameter: CLss/F of SOF, VEL, and VOX
Description: CLss/F is defined as the apparent steady state oral clearance following administration of the drug.
Time Frame: as for outcome 20
Population: Participants in the PK Analysis Set who were enrolled in Part B and received NGM+ SOV/VEL/VOX + VOX were analyzed.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15
mL/h
  SOF | 218383.1 (53265.75)
  VEL | 12757.3 (2673.70)
  VOX | 56071.5 (15234.72)

27. Secondary Outcome: PK Parameter: t1/2 of SOF, SOF Metabolites (GS-566500 and GS-331007), VEL, and VOX
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: as for outcome 20
Population: Participants in the PK Analysis Set who were enrolled in Part B and received NGM+ SOV/VEL/VOX + VOX were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Part B: NGM/EE + SOF/VEL/VOX + VOX
Number analyzed (Participants) | 15
hours
  SOF | 0.68 [0.45 to 0.81]
  GS-566500 | 2.70 [2.61 to 3.04]
  GS-331007 | 30.06 [24.96 to 75.66]
  VEL | 19.75 [15.46 to 24.92]
  VOX | 8.51 [7.56 to 13.55]

ADVERSE EVENTS:
Time Frame: First dose date up to the last dose date (maximum: 84 days) plus 10 days
Description: The Safety Analysis Set included all enrolled participants who took at least 1 dose of study drug.
Groups:
- Part A: NGM/EE: Participants received NGM 0.180 mg/0.215 mg/0.25 mg/ EE 0.025 mg tablet orally once daily for 1 cycle (cycle = 28 days).
- Part B: NGM/EE + SOF/VEL/VOX + VOX: Participants received NGM 0.180 mg/0.215 mg/0.25 mg/ EE 0.025 mg + sofosbuvir (SOF)/velpatasvir (VEL)/voxilaprevir (VOX) FDC 400/100/100 mg tablet + VOX 100 mg orally once daily for 2 cycles (cycle = 28 days).
Arm/Group | Part A: NGM/EE | Part B: NGM/EE + SOF/VEL/VOX + VOX
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 10/15 | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: NGM/EE (N=15) | Part B: NGM/EE + SOF/VEL/VOX + VOX (N=15)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Flatulence (Gastrointestinal disorders) | 0 | 2
Gingival ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 9
Vomiting (Gastrointestinal disorders) | 0 | 3
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 3
Hypersensitivity (Immune system disorders) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 6 | 6
Presyncope (Nervous system disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years